CLINICAL TRIAL: NCT03818022
Title: Effectiveness of Preoperative Cryoneurolysis (Iovera) for Postoperative Pain Control in Total Knee Arthroplasty
Brief Title: Pain Control With Pre-operative Cryoneurolysis Following TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost interest in study
Sponsor: Fondren Orthopedic Group L.L.P. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOH180
Record Dates: First submitted 2019-01-09; First posted 2019-01-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Osteo Arthritis Knee
Keywords: knee; joint replacement; total knee; cryoneurolysis; Iovera; TKA; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients receiving Cryoneurolysis (Iovera) prior to total knee arthroplasty
  Interventions: Procedure: Cryoneurolysis (Iovera)
- Control (No Intervention)

INTERVENTIONS:
Procedure: Cryoneurolysis (Iovera) — Cryoneurolysis performed by radiology department 1 week prior to total knee arthroplasty
  Arms: Experimental

SUMMARY:
The purpose of this study is to assess the potential benefit of preoperative cryoneurolysis in postoperative pain management of total knee arthroplasty patients over current pain management protocol.

DETAILED DESCRIPTION:
Cryoneurolysis, is a novel technique that can yield temporary blockade of superficial sensory nerves, generating immediate and meaningful relief of pain.The technique generates an axonotmesis of the targeted peripheral nerves by percutaneously applying low temperatures (-100 °C to -20 °C). Wallerian degeneration is produced whereby the axons and the myelin sheath are damaged but the endoneurium, perineurium and epineurium remain intact. Therefore, permanent damage to the nerve is avoided as it retains its regenerative properties. With regards to the knee, the infrapatellar branch of the saphenous nerve (IPBSN), a sensory branch serving both the inferior and anterior portion of the knee capsule and the antero-medial skin of the knee is the prime target for the procedure.

Your participation in this study requires that you allow the radiology department of Texas Orthopedic Hospital to administer Cryoneurolysis using the Iovera device with the functional smart tip approximately 1 week prior to total knee arthroplasty surgery. A highly localized cold zone is created via the Joule-Thompson effect as nitrous oxide enters the needles. Nothing is injected into the body and the nitrous oxide gas is vented safely out of the handpiece. Cryoneurolysis is administered following local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* any patient scheduled for primary total knee arthroplasty(TKA)

Exclusion Criteria:

* Bilateral TKA (patients routinely receive spinal anesthesia)
* Minors
* Patients reporting a history of Raynaud's disease
* Patients with an open and/or infected wound on surgical knee
* Patients who are taking opioids during the pre-operative period due to knee pain
* Patients who cannot return for the cryoneurolysis treatment 7 days prior to surgery or post-operative clinical visits
* Patients whose insurance would deny payment for the cryoneurolysis treatment
* Pregnant patients
* Patients unable to speak and read English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Veterans Rand-12 (VR-12) | up to 3 months
  VR-12 is a 12 item questionnaire that measures health related quality of life. Scores range from 0 to 100 with 50 being an average score and higher scores representing better health related quality of life.
Knee Injury and Osteoarthritis Outcomes Survey (KOOS Jr) | up to 3 months
  KOOS Jr. is a short questionnaire that evaluates knee pain and function. Scores range from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.

SECONDARY OUTCOMES:
Number of subject with an adverse effect from treatment | up to 3 months
  Any complication during treatment will be recorded.
Range of motion | up to 3 months
  During clinical office visits, your ability to bend and straighten your knee will be recorded.
Knee function | up to 3 months
  During clinical office visits, your ability to perform daily activities with regards to your knee will be recorded.
Knee swelling | up to 3 months
  The amount of swelling in your knee will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondren Orthopedic Group, L.L.P., Houston, Texas, United States